CLINICAL TRIAL: NCT05932043
Title: What Can I do for my Low Back Pain? The Work In Progress Questionnaire!
Brief Title: Development of the Work In Progress Questionnaire
Acronym: WIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Institute of Behavioral Medicines (Other)
Responsible Party: Principal Investigator, Barbara Rocca, Dr, International Institute of Behavioral Medicines
Other Study IDs: 2023-001
Record Dates: First submitted 2023-06-16; First posted 2023-07-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: outcome measures; commitment; people; psychology; behavioural medicine
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: This is a non-interventional study — None (this is a non-interventional study)

SUMMARY:
The aim of this study is to describe the development of the Work In Progress questionnaire, a tool designed to evaluate commitment in persons, and its psychometric validation process in the context of low back pain.

DETAILED DESCRIPTION:
The study design is cross-sectional.

The following methodology will be applied as for the development of the Work In Progress questionnaire (WIP), a tool designed to evaluate commitment in persons, and its psychometric validation:

1. item generation and selection: the first defines the content of an index and ensures the most important topics are well-thought-out. The second eliminates redundant items, and decreases the number to a total that is feasible to administer while ensuring the scale measures the construct of interest.
2. psychometric analysis: exploratory factor analysis (Cattel Scree Test, Varimax Rotation), reliability (internal consistency by Cronbach's alpha, test-retest reliability by Intraclass Correlation Coefficient 2.1), Measurement error (calculated by multiplying the standard error of measurement (SEM) by the z-score associated with the desired level of confidence (95%, in our case) and the square root of 2), and construct validity by hypothesis testing the correlations (Pearson r) with related measures (Pain Catastrophizing Scale, Oswestry Disability Scale, Numerical pain Rating Scale).

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain
* adult age
* reading/speaking Italian.

Exclusion Criteria:

* systemic illness, mental deficits, recent cerebrovascular accidents or myocardial infarctions, chronic lung or renal diseases;
* refusal to adhere.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with non-specific low back pain. For full description od the condition, please see the definition provided within the references list (Chiarotto A et al).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
WIP questionnaire | At the moment of the questionnaire administration
  Work In Progress questionnaire; score varying from 0 to 30, with higher scores indicating greater commitment
WIP questionnaire | After 7-10 days later the first assessment (please, see above) as concerns test-retest assessment reliability.
  Work In Progress questionnaire; score varying from 0 to 30, with higher scores indicating greater commitment

SECONDARY OUTCOMES:
PCS | At the moment of the questionnaire administration
  Pain Catastrophizing Scale; score varying from 0 to 52, with higher scores indicating greater catastrophizing
ODI | At the moment of the questionnaire administration
  Oswestry Disability Index; score varying from 0 to 50, with higher scores indicating greater disability
pain NRS | At the moment of the questionnaire administration
  Numerical pain Rating Scale; score varying from 0 to 10, with higher scores indicating greater pain intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Rocca, Calosso, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guyatt GH, Bombardier C, Tugwell PX. Measuring disease-specific quality of life in clinical trials. CMAJ. 1986 Apr 15;134(8):889-95. PMID 3955482
- [Result] Collins D. Pretesting survey instruments: an overview of cognitive methods. Qual Life Res. 2003 May;12(3):229-38. doi: 10.1023/a:1023254226592. PMID 12769135
- [Result] de Vet HCW, Terwee CB, Mokkink LB, et al. Measurement in medicine. A practical guide. Cambridge: Cambridge University Press, 2011
- [Result] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Result] Chiarotto A, Koes BW. Nonspecific Low Back Pain. N Engl J Med. 2022 May 5;386(18):1732-1740. doi: 10.1056/NEJMcp2032396. No abstract available. PMID 35507483
- [Result] Hayes SC. Get out of your mind and into your life: The new acceptance and commitment therapy. New Harbinger Publications; 2005 Nov 1.
- [Result] Sullivan MJ, Bishop SR, & Pivik J. The Pain Catastrophizing Scale: Development and validation. Psychol Assess 1995;7:524-532
- [Result] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Result] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508